CLINICAL TRIAL: NCT04233177
Title: Influence of Anesthesia, Pneumoperitoneum, and Patient Position on Common Carotid Artery Blood Flow During Laparoscopic Gynecology Operation
Brief Title: The Effect of Trendelenburg Position on CCA Blood Flow
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: CCA-BF
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Perfusion; Perioperative/Postoperative Complications
Keywords: Common carotid artery; Trendelenburg; Pneumoperitoneum; Blood flow
MeSH Terms: conditions — Postoperative Complications; Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will evaluate the change of the common carotid artery blood flow according to patient's position and penumoperitoneum.

DETAILED DESCRIPTION:
The study will include 20 patients undergoing gynecological surgery. The common carotid artery blood flow will be measured using Doppler US during the following conditions; supine position before induction of anesthesia, supine position immediately after induction of anesthesia, supine position with penumoperitoneum, head-down position with or without pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I,II
* patients undergoing gynecology surgery under trendelenburg position
* Age ranges from 20 to 70

Exclusion Criteria:

* BMI > 32
* Pregnancy
* Patients who did not agree to study
* Patients with allergies to the drugs used in this study
* Patients with anatomical variations or lesions in cervical or cranial vascular portion
* Patients with arrhythmia that may alter patient's cardiac output(e.g. artrial fibrillation)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing gynecology surgery under trendelenburg position
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Change of the common carotid artery blood flow velocity | 1) baseline, 2) Immediately after induction of anesthesia, 3) immediately after pneumoperitoneum, 4) immediately after Trendelenburg position with penumoperitoneum, 5) Immediately after desufflation in Trendelenburg position
  Common carotid artery blood flow velocity is measured using Doppler US

SECONDARY OUTCOMES:
Change of the common carotid artery beat volume | 1) baseline, 2) Immediately after induction of anesthesia, 3) immediately after pneumoperitoneum, 4) immediately after Trendelenburg position with penumoperitoneum, 5) Immediately after desufflation in Trendelenburg position
  Common carotid artery beat volume was calculated from median common carotid artery beat velocity and vessel diameter
Change of the common carotid artery diameter | 1) baseline, 2) Immediately after induction of anesthesia, 3) immediately after pneumoperitoneum, 4) immediately after Trendelenburg position with penumoperitoneum, 5) Immediately after desufflation in Trendelenburg position
  Common carotid artery diameter is obtained using US
Change of mean arterial blood pressure | 1) baseline, 2) Immediately after induction of anesthesia, 3) immediately after pneumoperitoneum, 4) immediately after Trendelenburg position with penumoperitoneum, 5) Immediately after desufflation in Trendelenburg position
  Mean arterial pressure is obtained concurrently with common carotid artery blood flow velocity measurements
Change of cardiac output | 1) baseline, 2) Immediately after induction of anesthesia, 3) immediately after pneumoperitoneum, 4) immediately after Trendelenburg position with penumoperitoneum, 5) Immediately after desufflation in Trendelenburg position
  Cardiac output was obtained using FloTrac(EdwardLifescience, USA)
Change of peak inspiration airway pressure | 1) baseline, 2) Immediately after induction of anesthesia, 3) immediately after pneumoperitoneum, 4) immediately after Trendelenburg position with penumoperitoneum, 5) Immediately after desufflation in Trendelenburg position
  Peak inspiratory airway pressure is obtained using the ventilator system

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon HK, Bae H, Yoo S, Kim YW, Bae J, Park SK, Kim H, Lim YJ, Kim JT. Relationships between common carotid artery blood flow and anesthesia, pneumoperitoneum, and head-down tilt position: a linear mixed-effect analysis. J Clin Monit Comput. 2023 Apr;37(2):669-677. doi: 10.1007/s10877-022-00940-z. Epub 2022 Dec 4. PMID 36463542